CLINICAL TRIAL: NCT05179720
Title: The Application Research of Ultrasound Guided Puncture Stent Assisted Transperineal Prostate Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CSZ02
Record Dates: First submitted 2021-12-01; First posted 2022-01-05 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients in the experimental group used a puncture stent to assist transperineal prostate biopsy.
Who Masked: Outcomes Assessor
Masking Description: Randomly assign patient groups according to the random number method.The biopsy sample inspector does not know the patient's biopsy method
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- puncture stent-assisted transperineal prostate biopsy (Experimental): This group of patients underwent puncture stent-assisted transperineal prostate biopsy.
  Interventions: Other: puncture stent-assisted transperineal prostate biopsy
- transperineal free-hand biopsy (Active Comparator): This group of patients underwent perineal free-hand biopsy
  Interventions: Other: puncture stent-assisted transperineal prostate biopsy

INTERVENTIONS:
Other: puncture stent-assisted transperineal prostate biopsy — Patients in the experimental group used a puncture stent to assist transperineal prostate biopsy

SUMMARY:
This study is a multi-center prospective study. Patients who meet the indications for prostate biopsy were included in this study.The study was randomly divided into two groups, one group was transperineal free-hand biopsy; the other group was puncture stent-assisted transperineal prostate biopsy. Exploring the positive rate of puncture stent-assisted transperineal prostate biopsy

DETAILED DESCRIPTION:
This study is a multi-center prospective study. Patients who meet the indications for prostate biopsy were included in this study.The study was randomly divided into two groups, one group was transperineal free-hand biopsy; the other group was puncture stent-assisted transperineal prostate biopsy. Exploring the positive rate of puncture stent-assisted transperineal prostate biopsy 560 patients were enrolled. The main result is the positive rate of biopsy: including the detection rate of clinically meaningful prostate cancer and the detection rate of clinically insignificant prostate cancer.Secondary results include: (1)Biopsy complications include (infection, bleeding, etc.).(2)Pain score of biopsy patients (NRS score).(3) Biopsy time

ELIGIBILITY:
Inclusion Criteria:

Suspected prostate cancer patients Can tolerate prostate puncture

Exclusion Criteria:

Symptomatic acute or chronic inflammation of the prostate Patients with other cancers

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
positive rate of biopsy | 1 year
  Including the detection rate of clinically meaningful prostate cancer and the detection rate of clinically insignificant prostate cancer

SECONDARY OUTCOMES:
Biopsy complications include (infection, bleeding, etc.) | 1 year
  Biopsy complications include (infection, bleeding, etc.)
Pain score of biopsy patients (NRS score) | 1 year
  Pain score of biopsy patients (NRS score)
Biopsy time | 1 year
  Biopsy time

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital, Jinan, Shandong, China